CLINICAL TRIAL: NCT05099822
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-center, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of CC-97489 in Healthy Adult Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CC-97489 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CC-97489-CP-001; 2019-003458-10 (EudraCT Number)
Record Dates: First submitted 2021-09-09; First posted 2021-10-29 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
Keywords: CC-97489; Healthy Adult; Phase1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of CC-97489 (Experimental)
  Interventions: Drug: CC-97489
- Administration of Placebo (Experimental)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-97489 — Specified dose on specified days
  Other Names: BMS-986368
  Arms: Administration of CC-97489
Other: Placebo — Specified dose on specified days
  Arms: Administration of Placebo

SUMMARY:
This study aims to evaluate the safety, tolerability, of CC-97489

ELIGIBILITY:
Inclusion Criteria:

* In good health, as determined by the investigator based on past medical history, physical examination, vital signs and clinical laboratory safety tests at screening.
* Body mass index (BMI) ≥ 18 and ≤ 33 kg/m^2, inclusive. BMI = weight (kg)/(height [m])^2

Exclusion Criteria:

• Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, echocardiogram (ECG), or clinical laboratory determinations beyond what is consistent with healthy participants

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 28 days after the last dose
Incidence of Serious Adverse Events (SAEs) | 28 days after the last dose
Number of participants with clinically significant changes in electrocardiogram parameters | Day 21
Incidence of clinically significant changes in vital signs: Body temperature | Day 21
Incidence of clinically significant changes in vital signs: Respiratory rate | Day 21
Incidence of clinically significant changes in vital signs: Blood pressure | Day 21
Incidence of clinically significant changes in vital signs: Heart rate | Day 21
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Day 18
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Day 18
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Day 18

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum observed plasma concentration (Cmax) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Minimum plasma drug concentration (Cmin) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Time to maximum observed plasma concentration (Tmax) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Area under the plasma concentration (AUC)-time curve from time zero extrapolated to infinity (AUC0-∞) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Area under the plasma concentration-time curve from time zero to time t, where t is the time point of the last measurable concentration (AUC0-t) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Area under the plasma concentration-time curve from time zero to 24 hours postdose (AUC0-24) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Area under the plasma concentration-time curve from time zero to tau (τ) where τ is the dosing interval (AUC0- 0-τ) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Terminal elimination half-life in plasma (t½,z) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Apparent total plasma clearance when dosed orally (CL/F) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Apparent total volume of distribution when dosed orally (Vz/F) | Up to 96 hours after the last dose of study drug
Pharmacokinetics - Ratio of accumulation based on Day 1 and Day 14 AUC0- 0-τ and Cmax, as appropriate (Rac) | Up to 96 hours after the last dose of study drug
Pharmacodynamics - Evaluation of monoacylglycerol lipase (MGLL) enzymatic inhibition by CC-97489 in peripheral blood mononuclear cells (PBMCs) | Up to 168 hours after the last dose of study drug
Pharmacodynamics: Peripheral blood mononuclear cell (PBMC) fatty acid amide hydrolase (FAAH) inhibition | Up to 168 hours after the last dose of study drug
Pharmacodynamics - Measurement of : plasma and whole-blood anandamide (AEA) levels | Up to 168 hours after the last dose of study drug
Pharmacodynamics - Measurement of plasma and whole-blood 2-arachidonoylglycerol (2-AG) levels | Up to 168 hours after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 001, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com